CLINICAL TRIAL: NCT01489410
Title: Prospective Study Comparing Lipiodol Plus Ethanol Solution Compared With Drug-Eluting Beads for Trans-arterial Chemoembolization of Liver in Treatment of Hepatocellular Carcinoma
Brief Title: Comparing Lipiodol/Ethanol With Drug-eluting Beads (DEB) for Hepatocellular Carcinoma
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient staff
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2011LS117
Record Dates: First submitted 2011-12-06; First posted 2011-12-09 (Estimated); Last update posted 2017-08-31 (Actual); Status verified 2017-08

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Drug-Eluting Beads with Doxorubicin (Active Comparator): Drug-Eluting Beads (DEB) with Doxorubicin is administered via beads that release it to the liver through a groin puncture site and delivered via catheter through the vessels that feed the liver.
  Interventions: Drug: Drug-Eluting Beads (DEB) with Doxorubicin
- Lipiodol Ethanol Mixture (LEM) (Active Comparator): Lipiodol Ethanol Mixture (LEM) is administered to the liver through a groin puncture site and delivered via catheter through the vessels that feed the liver.
  Interventions: Drug: Lipiodol Ethanol Mixture

INTERVENTIONS:
Drug: Drug-Eluting Beads (DEB) with Doxorubicin — One treatment of Drug-Eluting Beads (DEB) with Doxorubicin administered to the liver through a groin puncture site and delivered through the vessels that feed the liver (per standard of care).
  Other Names: Doxorubicin
  Arms: Drug-Eluting Beads with Doxorubicin
Drug: Lipiodol Ethanol Mixture — One treatment of Lipiodol Ethanol Mixture (LEM) is administered to the liver through a groin puncture site and delivered through the vessels that feed the liver (per standard of care).
  Other Names: LEM
  Arms: Lipiodol Ethanol Mixture (LEM)

SUMMARY:
Chemoembolization of hepatocellular carcinoma lesions is an accepted and frequently used method for the palliative or curative treatment of these lesions. These attempts are being made to make these patients a better candidate for liver transplant or to provide palliation for their condition.

DETAILED DESCRIPTION:
This is a randomized prospective study with two arms, Drug-Eluting Beads with doxorubicin (DEB) and lipiodol ethanol mixture (LEM), with the goal to show non-inferiority of LEM, which if true will facilitate a simple alternative to DEBs. Patients will be randomized to one arm of the study and will remain in that arm if they need to have more embolization in the future. Both of the mentioned methods (DEB and LEM) fall within the standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Child-Pugh class A or B
* Biopsy proven HCC or hypervascular mass per European Association for the Study of the Liver (EASL) criteria
* Patient not a candidate for surgical resection or percutaneous ablation
* age > 18 years old and able to consent

Exclusion Criteria:

* Child-Pugh class C
* Model for End-Stage Liver Disease (MELD) score >16
* Extrahepatic disease
* Bilateral or main portal vein thrombus
* Total bilirubin > 2.2
* Serum albumin < 2.6
* Life expectancy < 2 months
* Uncorrected INR > 2
* Eastern Cooperative Oncology Group (ECOG) status > 2
* Tumor burden > 50% liver volume
* Hepatofugal portal venous flow

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-10; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Number of Patients with Post-Embolization Syndrome | Week 6 Post Intervention
  Count of patients with post-embolizaation syndrome reported which includes fatigue, anorexia, nausea, fever.

SECONDARY OUTCOMES:
Patients with Encephalopathy After Embolization | Week 6 Post Intervention
  Count of patients who had encephalopathy after embolization.
Changes in Quality of Life | Baseline and Week 6 After Intervention
  Changes (noted as a score of 0 [not at all] to 4 [very much]; total score ranges from 1-180) in the different aspects of the Functional Assessment of Cancer Therapy-Hepatobiliary (FACT-Hep) quality of life questionnaire (a 45-item self-report instrument designed to measure health-related quality of life in patients with hepatobiliary cancers).
Comparison of Liver Function Tests Results | Day 0 and Week 6 Post Intervention
  List of results for alpha-fetoprotein (AFP), albumin (Alb), alanine transaminase (ALT), aspartate aminotransferase (AST), alkaline phosphatase (ALKP), blood urea nitrogen (BUN), creatinine (Cr), glomerular filtration rate (GFR), Bilirubin (T, D), platelets (Plt), international normalized ratio (INR - prothrombin time), Child-Pugh score.
Imaging Response | Week 6 Post Intervention
  Determined by European Association for the Study of the Liver (EASL) criteria a set of non-invasive criteria for HCC in cirrhotic patients. The diagnosis is established if two imaging modalities (US, CT, magnetic resonance imaging (MRI)) show a coincidental nodule with arterial hypervascularization regardless of AFP levels, or if a single modality shows a lesion when the AFP levels are more than 400 ng/ml. Histologic diagnosis is required if the patient is non-cirrhotic or if the lesions are smaller than 2 cm.
Number of Patients with Successful Liver Transplant | Week 6 After Intervention
Overall Survival | Week 6 After Intervention
  Determined by date of death or date censored.

CONTACTS AND LOCATIONS:
Overall Officials: Erik Cressman, M.D., Principal Investigator — Masonic Cancer Center, University of Minnesota
Locations (1):
- Masonic Cancer Center, University of Minnesota, Minneapolis, Minnesota, United States